CLINICAL TRIAL: NCT07252973
Title: Sustainable Anaesthesia Practices in EUROPE
Brief Title: Sustainable Anaesthesia Practices in EUROPE - a Prospective International Cohort Study
Acronym: SUSTAIN-EUROPE
Status: Not yet recruiting | Type: Observational
Sponsor: European Society of Anaesthesiology (Other)
Responsible Party: Sponsor
Other Study IDs: CTN_SUSTAIN-EUROPE
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Anaesthesia Conduction; Paediatric and Adult Patients; Carbon Footprint in Anesthetic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Anaesthesia technique — Observation of type of anaesthesia used in Europe

SUMMARY:
In response to the climate crises, Societies of Anaesthesiology around the globe call for action to reduce the carbon footprint of daily clinical work. They recommend the use of regional and total intravenous anaesthesia, and for inhalational anaesthesia cases, the use of sevoflurane with low fresh gas flow (FGF < 0.5 lpm) settings. Surprisingly, the type of anaesthesia and ventilation settings commonly used remain largely unknown. This pragmatic observational cross-sectional assessment at all anaesthesia workstations in participating European hospitals in daily routine aims to evaluate anaesthesia practices in the paediatric and adult patient population.

ELIGIBILITY:
Inclusion Criteria:

* All patients receiving any form of anaesthesia care-whether general or regional anaesthesia, monitored sedation, or monitoring only-from an anaesthetist at an anaesthesia workstation in participating European hospitals during the selected data-collection recruitment period

Exclusion Criteria:

* Patients (or legal guardians) who decline consent and patients for whom valid informed consent cannot be obtained due to language barriers or other factors preventing adequate information and understanding.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: SUSTAIN-EUROPE is designed to close the knowledge gap on contemporary anaesthesia practices in both adult and paediatric populations
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Type of anaesthesia (inhalational and intravenous general anaesthesia, regional anaesthesia, sedation, combinations, monitoring only) | 5-60 min after the skin incision
  The type of anaesthesia (inhalational and intravenous general anaesthesia, regional anaesthesia, sedation, combinations, or monitoring only) will be recorded by a trained team member collecting data perioperatively 5-60 minutes after skin incision or start of procedure, respectively. In the event that the anaesthetic approach changes intraoperatively, only the technique recorded at that time point will be used for analysis. Any local anaesthetic infiltration performed by the anaesthetist will be classified as regional anaesthesia, whereas if the surgeon alone administers local anaesthetic, this will not be classified by regional anaesthesia.

IPD SHARING:
Plan to Share IPD: No